CLINICAL TRIAL: NCT02809898
Title: The Role of ctDNA and PBMC as Biomarkers in Diagnostic, Efficacy Monitoring and Prognostic Evaluation of Biliary Tract Cancer
Brief Title: The Role of ctDNA and PBMC in Treatment of Biliary Tract Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Huadong Hospital (Other); Shanghai Changzheng Hospital (Other); Yangpu District Central Hospital Affiliated to Tongji University (Other)
Responsible Party: Sponsor
Other Study IDs: cfDNA-GCCC
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Biliary Tract Neoplasms
Keywords: Biomarkers, Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms; Neoplasms | interventions — Surgical Procedures, Operative; Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: surgery or biopsy — Do radical surgery or biopsy to obtain a pathological result

SUMMARY:
Our study aims to evaluate the role of ct-DNA and PBMC as biomarkers in the treatment of biliary tract cancer.

DETAILED DESCRIPTION:
Biliary cancer ranked fifth in all gastrointestinal malignant cancer. Epidemiological surveys showed a significant increasing trend in recent years. How can make an early diagnosis of bile duct cancer as well as prognostic evaluation and efficacy monitoring, has become the hotspot. "liquid biopsy", which is meant to detect cancers by sequencing the DNA in a few drops of a person's blood. It may detect cancers early, even before symptoms arise, when there is just a few cells in the blood circulation.

cf-DNA in cancer patients often bears similar genetic and epigenetic features to the related tumor DNA. There is evidence that some of the cf-DNA originates from tumoral tissue. This, and the fact that cf-DNA can easily be isolated from the circulation and other body fluids of patients, makes it a promising candidate as a non-invasive biomarker of cancer. And we call the cf-DNA of tumor as ct-DNA.

Peripheral blood mononuclear cells (PBMC) is any peripheral blood cell having a round nucleus. These cells can be extracted from whole blood using ficoll, a hydrophilic polysaccharide. PBMC contains genetic material of tumor and may be applied as a biomarker.

This study aims to evaluate the role of ct-DNA and PBMC as biomarkers in the treatment of biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected biliary tract cancer
* Age from 18 - 70 years
* No serious organic and mental illness;

Exclusion Criteria:

* Pregnancy
* No pathologic result
* Suffering other malignancies at the same time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected biliary tract cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pathological diagnosis of gallbladder polyps （Cholesterol / Adenoma / Others） | intraoperative
  Sensitivity and specificity

SECONDARY OUTCOMES:
Tumor status （worse/ maintain/ better） | 3 years
  the level of ct-DNA compared with the tumor burden

CONTACTS AND LOCATIONS:
Overall Officials: Tao Chen, M.D., Principal Investigator — Department of Biliary-pancreatic Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (4):
- China (4):
  - Huadong Hospital, Shanghai
  - Shanghai Yangpu district central hospital, Shanghai
  - Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai
  - Shanghai Changzheng Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided